CLINICAL TRIAL: NCT02491307
Title: Ginger.io Behavioral Health Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Community Health Center, Inc. (Industry)
Collaborators: Ginger.io (Industry); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1059
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Anxiety; Depression; Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Anxiety Disorders; Depression; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginger.io Application Users (Experimental): This cohort is comprised of individuals that 1) are English-speaking; 2) possess an Android or iOS smartphone; 3) have a diagnosis for anxiety, depression, and/or bipolar disorder; and 4) are active behavioral health patients at any of the four CHCI clinic sites (New London, New Britain, Middletown, or Meriden) where behavioral health providers are using the Ginger.io app with their patients. These patients receive the Ginger.io smartphone application for daily use.
  Interventions: Other: Ginger.io Smartphone Application
- Non-application users (No Intervention): This cohort is comprised of individuals that 1) are English-speaking; 2) possess an Android or iOS smartphone; 3) have anxiety, depression, and/or bipolar disorder; and 4) are patient of a behavioral health clinician that is providing paper surveys to patients in clinic. They do not receive the Ginger.io smartphone application.

INTERVENTIONS:
Other: Ginger.io Smartphone Application — Daily use of the Ginger.io smartphone application
  Arms: Ginger.io Application Users

SUMMARY:
This Study will evaluate the impact of a smartphone-based platform on a range of outcomes for medically-underserved patients with mood disorders (e.g. depression, anxiety, bipolar) cared for in a large statewide community health center. The primary goal of the Study is to reduce emergency room (ER) visits, hospitalizations, and to look at changes in service utilization by using the Ginger.io platform to enhance communication between behavioral health providers and their patients, increasing the early detection of exacerbations in mood disorders (e.g. depression, anxiety, bipolar) and proactive outreach. The secondary goal is to improve clinical & behavioral health outcomes.

DETAILED DESCRIPTION:
Procedures involved in the Human Research Overview: The investigators will use a quasi-experimental study with a pre-post intervention design to evaluate the usability, feasibility, acceptability, and potential utility of a smartphone app to improve patient-behavioral health provider communication and care for patients with mood disorders (e.g. depression, anxiety, bipolar). The smartphone app will collect patient smartphone interaction data and survey data from patients on their health and functioning including mood, depression, and anxiety levels. At various points during the study, patients will be surveyed about their experience using the smartphone application, Ginger.io.

All behavioral health providers at Community Health Center, Inc. (CHCI) who are using the app with their patients will be granted access to a secured, password-protected, web-based dashboard that will collect and display information related to patients' health and behavior. The research assistant and behavioral health providers will use the web-based dashboard to monitor patient activation and survey completion, and the behavioral health provider will use it to proactively reach out to patients and aid in discussions with the patient about the care he/she receives at CHCI. At various points during the study, behavioral health providers will be surveyed about their experience using the secured, password-protected web-based provider dashboard.

Behavioral health providers at multiple CHCI sites will be using this app with their patients as part of their care. From the pool of Ginger.io existing users, about 500 patients will sign written informed consent and join the research study. These patients will provide survey information that will be used in the research study. Comparison data will also be gathered from CHCI's electronic health record and via the completion of paper surveys for approximately 100 patients that sign written informed consent and who are receiving routine behavioral health care at CHCI but are not using the Ginger.io app. Baseline data on the patient's depression, bipolar and anxiety will be collected the first time using the Ginger.io app or filling out paper forms in control clinics.

Intervention patients will be asked to use the Ginger.io smartphone app for a minimum of 6 months, to answer depression, anxiety and mood questions. The Ginger.io app may also be used by patients on a less frequent (e.g. weekly, biweekly, or monthly) basis to answer more detailed surveys like the self-report hospitalization or Patient Health Questionnaire (PHQ-9), which collects data on depression. These daily and weekly assessments of patient mood, depression and anxiety, including data on the patient's mobility and communication, will be collected by the Ginger.io smartphone application, and available 24/7 in the dashboard, so that the dashboard monitor can take appropriate action (or should they choose, the behavioral health clinician could view as well at monthly visits). Most importantly, behavioral health providers will be performing proactive outreach to patients that are identified by alerts as being at higher likelihood of mood disorder irregularities. These alerts are powered by patient survey responses and smartphone passive behavioral changes.

Intervention Description:

Patient Data Collected Using the Ginger.io Smartphone Application:

Patients who are referred to the study by a participating behavioral health provider or are recruited via phone, email, etc. provide data for inclusion in the research study will be current users of the Ginger.io smartphone application that is available free of charge and will receive instruction on how to download and use the app if applicable. Once the app is installed on their phone, patients will receive prompts on their smartphone to complete assessments. The Ginger.io application will also collect data passively on the patient's levels of communication and mobility while using their smartphone. The patient will not be required to complete an assessment of communication and mobility - once the application is installed on the patient's smartphone, it will collect this data automatically. Patients will have the ability and option to turn these features off if that is their preference. Patients will be asked to use the Ginger.io application for at least six consecutive months. Communication and mobility data will also be collected by the application for the duration of the patient's participation in the study. Patients will also be asked to complete brief patient surveys about their experience with using the Ginger.io app. The data collection period will begin on the day of app download, but this data will not be examined for the purposes of this study until a patient has signed written informed consent documentation. When downloading the Ginger.io app, patients indicate their consent (or not) to allow the app to capture passive motion, mobility, and communication data. If the patient has allowed the Ginger.io app to capture this data, passive motion and mobility data will be used by the patient's behavioral health provider to supplement between-visit information provided by the patient while completing surveys. The data will also be used by CHCI and Ginger.io to refine and improve the threshold that triggers an alert that is generated by the Ginger.io app and sent to the CHCI behavioral health provider when it is suspected that the patient is experiencing exacerbated mental health symptoms. As mentioned, these features can be turned off by the patient. This passive data collection does not collect the content of calls or text messages and does not track the exact location of the patient (i.e. the patient went to a specific restaurant or store). It simply measures volumes of contact and amount of movement to attempt to identify deviations from normal (i.e. a patient no longer calls or texts anyone, a patient doesn't leave home for several days, a patient is using their phone in the middle of the night) to detect exacerbations of their mood disorder.

Alerts Triggered by Patient Responses to Ginger.io Survey Question Assessments:

When a patient's mood scores and activity exceed thresholds set by a predetermined Ginger.io algorithm, the Ginger.io app creates an alert. Alerts generated by the Ginger.io system will be relayed to behavioral health providers via the provider dashboard. The behavioral health provider will decide how best to respond, e.g. by contacting the patient or having a nurse or medical assistant contact the patient. Behavioral health providers will be asked to check for alerts at least once each business day. They will not be required to check on weekends or days off. A research assistant will have administrative access to all dashboards to ensure that behavioral health providers are checking and resolving alerts as they are received and that no alert goes unaddressed.

If a patient is completing surveys in a manner than indicates an emergency, the app will deploy a screen that informs that patient that they should seek help and presents them with contact information for the Suicide Hotline. Additionally, the written informed consent document that the patients will have a copy of will direct them for how to get after-hours help through CHCI and to call the Suicide Hotline or 911 in case of an emergency.

Patient and Behavioral Health Provider Review of Patients' Ginger.io Data:

While the main intervention is alert-enabled outreach, participating patients and their behavioral health providers will have the opportunity to review the patient's data should they desire, presented in graphical form in the dashboard. This summary will provide a longitudinal view of the patient's responses to questions about their health (including depression, bipolar and anxiety). Patients and behavioral health providers will be able to review these results together at behavioral health office visits and use them to inform their discussion about the patient's care experience, the efficacy of the patient's treatment regimen, and whether to modify the patient's treatment plan. Monthly during the study, behavioral health providers will be surveyed using Survey Monkey about their experience using the secured, password-protected web-based provider dashboard.

Periodic Delivery of Health Tips and Coping Strategies for Depression & Anxiety & Bipolar In addition to surveys, the Ginger.io app delivers periodic health tips. The tips are evidence-based, created by professional psychologists, and offer light-weight practical means for patients to cope with bipolar, depression & anxiety.

Data management Electronic Health Record Data: CHCI has an electronic health record system which includes all patient health records. The present study will use data elements from the system, including primary care performance measures, chart review data, pharmacy prescribing data, lab data and utilization data (outpatient visits, urgent visits). For each patient, an index date will be defined - for patients in the intervention group, the date will be the app activation date; for patients in the control group it will be a comparable visit date. Electronic health record data will be extracted for 6-months before and after the index date for each patient.

In addition to these data elements, the investigators will also analyze the survey data collected via the Ginger.io app.

The following are measures to be obtained by the research team:

1. Behavioral health provider measures:

   a. Monthly behavioral health provider surveys
2. Patient Measures:

   1. Bidaily depression, mood & anxiety
   2. Substance abuse questions
   3. Weekly treatment adherence question
   4. Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder Screen (GAD-7) biweekly, alternating
   5. A drug/alcohol screen:Single Question Alcohol Screen (SQAS), Single Question Drug Screen (SQDS), Alcohol Use Disorder Identification Test (AUDIT-C), Drug Abuse Screening Test (DAST-10)
   6. Hospitalization surveys
   7. Monthly app satisfaction surveys
   8. Comprehensive data will be collected from eClinical Works (ECW) for participating patients, including demographic data, co-morbidity, behavioral health diagnoses, clinic utilization, and medication prescribed.

Withdrawal of subjects Patient subjects will be able to withdraw from the study at any time without penalty. Patients may be withdrawn from the study by research personnel if they lose access to their smartphones for an extended period of time during the study period or if they uninstall the Ginger.io smartphone application without re-installing it. Enrolled patient participants who are not completing daily and weekly surveys on a consistent basis may be contacted by a Research Assistant or Ginger.io and offered technical assistance with using the application, if needed. Patients who accept this assistance may meet in-person with a Research Assistant to relearn how to use the app, or to re-install it, if necessary. Patients will be eligible to receive additional technical assistance from Research Assistants at any point during their enrollment in the study. All patient data collected using Ginger.io between enrollment in the study and withdrawal from the study will be retained and analyzed by the research team at CHCI and by Ginger.io.

CHCI behavioral health provider subjects may withdraw from the study at any time without penalty. Behavioral health providers who are found to not be following protocol will be contacted by research staff to inquire why. When a provider withdraws from the study, his or her enrolled patients will be given the option to stop providing study data via the Ginger.io smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Experiencing mood disorders (e.g. depression, anxiety, bipolar) defined as a visit with a specified DSM-V code (295.7 Schizoaffective Disorder (Depressive type), 295.7 Schizoaffective Disorder (Bipolar type), 296.41 Bipolar I Current or most recent episode manic Mild, 296.42 Bipolar I Current or most recent episode manic mod, 296.43 Bipolar I Current or most recent episode manic sev, 296.44 Bipolar I Current or most recent episode manic w psychotic, 296.45 Bipolar I Current or most recent episode manic in partial remission, 296.46 Bipolar I Current or most recent episode manic in full remission, 296.40 Bipolar I Current or most recent episode unspecified, 296.40 Bipolar I Current or most recent episode hypomanic, 296.45 Bipolar I Current or most recent episode hypomanic in partial remission, 296.46 Bipolar I Current or most recent episode hypomanic in full remission, 296.40 Bipolar I Current or most recent episode hypomanic unspecified, 296.51Bipolar 1 Current or most recent episode depressed mild, 296.52 Bipolar 1 Current or most recent episode depressed mod, 296.53 Bipolar 1 Current or most recent episode depressed sev, 296.54 Bipolar 1 Current or most recent episode depressed w psychotic, 296.55 Bipolar 1 Current or most recent episode depressed in partial remission, 296.56 Bipolar 1 Current or most recent episode depressed in full remission, 296.50 Bipolar 1 Current or most recent episode depressed unspecified, 296.7 Bipolar 1 current or most recent episode unspecified, 296.89 Bipolar II, 301.13 Cyclothymic, 296.83 Bipolar due to Medical Condition, 296.89 Other Specified Bipolar, 296.80 Unspecified Bipolar, 296.99 Disruptive Mood Dysregulation disorder, 296.21 Major Depressive Disorder Single Episode Mild, 296.22 Major Depressive Disorder Single Episode mod, 296.23 Major Depressive Disorder Single Episode sev, 296.24 Major Depressive Disorder Single Episode w psychotic, 296.25 Major Depressive Disorder Single Episode in partial remission, 296.26 Major Depressive Disorder Single Episode in full remission, 296.20 Major Depressive Disorder Single Episode unspecified, 296.31 Major Depressive Disorder Recurrent Episode mild, 296.32 Major Depressive Disorder Recurrent Episode moderate, 296.33 Major Depressive Disorder Recurrent Episode severe, 296.34 Major Depressive Disorder Recurrent Episode w psychotic, 296.35 Major Depressive Disorder Recurrent Episode in partial remission, 296.36 Major Depressive Disorder Recurrent Episode in full remission, 296.30 unspecified, 300.4 Persistent Depressive Disorder (Dysthymia), 625.4 Premenstrual Dysphoric Disorder, 293.83 Depressive Disorder due to another medical condition, 311 Other specified depressive disorder, 311 Unspecified Depressive disorder, 309.21 Separation anxiety disorder, 300.29 Specific Phobia, 300.23 Social anxiety do, 300.01 Panic Disorder, 300.22 Agoraphobia, 300.02 GAD, 293.84 Anxiety do due to another med condition, 300.09 other specified anxiety do, 300.00 Uspecified Anxiety do, 309.0 Adjustment do with depressed mood, 309.24 Adjustment do with anxiety, 309.28 Adjustment do with mixed, 309.4 Adjustment do with w disturbance of emotions and conduct, 309.9 Adjustment do unspecified, 300.7 Illness anxiety disorder, 293.83 Mood do NOS, 296.9 Mood do unspecified, 291.89 alcohol inducted mood do, 292.84 amphetamine inducted mood do 292.84 cocaine inducted mood do, unspecified inducted mood do, 296.66 episodic mood dis unspecified, 296.64 Severe mixed bipolar do)
* Possessing a smartphone with either an Android or iOS platform
* Able to read and write in English
* Have a designated primary behavioral health care provider who is either using the app with their patients (intervention) or is issuing the surveys on paper in their clinic (control)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Emergecny room and hospitalization Data | 6 months
  Data on hospitalizations and ER visits will be collected for each enrolled patient over a 6 month time frame through an in-app question and/or as recorded in the patient's EHR
Service Utilization | 6 months
  Data on visits to CHCI during the patient's 6 month enrollment will be extracted from the EHR and examined for volume and type.

SECONDARY OUTCOMES:
Patient activation/self-management | 6 months
  Measured via the Ginger.io smartphone app
Patient perceived physical health status | 6 months
Patient perceived mental health status | 6 months
Patient satisfaction/connectedness | 6 months
  Measured via survey
Behavioral Health provider satisfaction | 6 months
  Behavioral health providers will be issued a brief survey once a month to share their experience using Ginger.io
Behavioral health provider effectiveness score | 6 months
Progress towards treatment goals | 6 months
  Examines care plan and progress towards goals as recorded in the patient's EHR

CONTACTS AND LOCATIONS:
Overall Officials: David Guggenheim, PsyD, Principal Investigator — Community Health Center, Inc.; Ilan Elson, PhD, Principal Investigator — Ginger.io
Locations (4):
- United States (4):
  - Community Health Center, Inc.-Meriden, Meriden, Connecticut
  - Community Health Center, Inc.- Middletown, Middletown, Connecticut
  - Community Health Center, Inc.-New Britain, New Britain, Connecticut
  - Community Health Center, Inc.-New London, New London, Connecticut